CLINICAL TRIAL: NCT05327686
Title: Randomized Phase II Stereotactic Ablative Radiation Therapy (SABR) for Metastatic Unresected Renal Cell Carcinoma (RCC) Receiving Immunotherapy (SAMURAI)
Brief Title: Testing the Addition of Stereotactic Radiation Therapy With Immune Therapy for the Treatment of Patients With Unresectable or Metastatic Renal Cell Cancer, SAMURAI Trial
Acronym: SAMURAI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU012; NCI-2022-02189 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU012 (Other: NRG Oncology); NRG-GU012 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — avelumab; Axitinib; Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; lenvatinib; Magnetic Resonance Spectroscopy; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (standard of care immunotherapy) (Active Comparator): Patients receive one of the following immunotherapy regimens per physician discretion: nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes every 3 weeks for 4 doses followed by nivolumab IV over 30 minutes every 2 or 4 weeks; pembrolizumab IV over 30 minutes every 3 or 6 weeks and axitinib PO BID; avelumab IV over 60 minutes every 2 weeks and axitinib PO BID; nivolumab IV over 30 minutes every 2 or 4 weeks and cabozantinib PO QD; OR pembrolizumab IV over 30 minutes every 3 or 6 weeks and lenvatinib PO QD. Treatment with immunotherapy continues in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI throughout the trial. Patients may also undergo a bone scan as clinically indicated and blood sample collection throughout the trial.
  Interventions: Biological: Avelumab; Drug: Axitinib; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib; Procedure: Computed Tomography; Biological: Ipilimumab; Drug: Lenvatinib; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Biological: Pembrolizumab
- Arm II (SABR, standard of care immunotherapy) (Experimental): Patients undergo SABR on 3 different days over 1-3 weeks and receive immunotherapy as in Arm I. Patients also undergo CT scan or MRI throughout the trial. Patients may also undergo a bone scan as clinically indicated and blood sample collection throughout the trial.
  Interventions: Biological: Avelumab; Drug: Axitinib; Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Cabozantinib; Procedure: Computed Tomography; Biological: Ipilimumab; Drug: Lenvatinib; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Biological: Pembrolizumab; Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Biological: Avelumab — Given IV
  Other Names: Bavencio; MSB 0010718C; MSB-0010718C; MSB0010718C
Drug: Axitinib — Given PO
  Other Names: AG 013736; AG-013736; AG013736; Inlyta
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Cabozantinib — Given PO
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Drug: Lenvatinib — Given PO
  Other Names: E 7080; E-7080; E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Radiation: Stereotactic Ablative Radiotherapy — 42 Gy in 3 fractions
  Other Names: SABER; SABR/SBRT
  Arms: Arm II (SABR, standard of care immunotherapy)

SUMMARY:
This phase II trial tests whether the addition of radiation to the primary tumor, typically given with stereotactic ablative radiation therapy (SABR), in combination with standard of care immunotherapy improves outcomes in patients with renal cell cancer that is not recommended for surgery and has spread from where it first started (primary site) to other places in the body (metastatic). Radiation therapy uses high energy photons to kill tumor cells and shrink tumors. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses of radiation over a shorter period and cause less damage to normal tissue. Immunotherapy with monoclonal antibodies, such as nivolumab, ipilimumab, avelumab, and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Axitinib, cabozantinib, and lenvatinib are in a class of medications called antiangiogenic agents. They work by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Giving SABR in combination with standard of care immunotherapy may help shrink or stabilize the cancer in patients with renal cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the addition of stereotactic ablative radiotherapy (SABR) to the primary tumor in combination with immunotherapy improves outcomes compared to immunotherapy alone in patients with metastatic, unresected, renal cell carcinoma (RCC). The primary endpoint is nephrectomy and radiographic progression-free survival (nrPFS) with progression determined as per iRECIST criteria.

SECONDARY OBJECTIVES:

I. To assess the safety, toxicity and tolerability of the two treatment strategies as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5 in each treatment arm.

II. To assess the objective response rate (ORR) by Immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) in each treatment arm.

III. Nephrectomy and radiographic progression-free survival excluding nephrectomies that were performed for non-protocol specified indications (nephrectomy and radiographic progression-free survival [nrPFS]2).

IV. Radiographic progression-free survival (rPFS). V. To assess overall survival (OS) in each treatment arm. VI. To assess the time to subsequent second-line therapy or death in each treatment arm.

VII. To assess the rate of cytoreductive nephrectomy in each treatment arm. VIII. To assess treatment-free survival in patients who discontinue therapy for reason other than radiographic disease progression.

IX. To assess the ORR by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and iRECIST in the primary renal mass.

EXPLORATORY OBJECTIVES:

I. To assess composite nrPFS in the predefined histological subgroups below:

Ia. Clear cell versus non-clear cell histology; Ib. International Metastatic RCC database consortium (IMDC) intermediate versus poor risk group; Ic. Systemic treatment with immunotherapy-immunotherapy combination versus immunotherapy-vascular endothelial growth factor (VEGF) targeted therapy combination; Id. Sarcomatoid versus non sarcomatoid variant. II. To identify prognostic and predictive biomarkers of response to SABR in the context of immunotherapy based treatment via assessment of tissue and blood based biomarkers.

III. To evaluate the abscopal effect of SABR with systemic therapy. IIIa. Compare ORR in non-irradiated target lesions in the control arm patients undergoing immunotherapy alone to the experimental arm undergoing SABR + immunotherapy.

IV. To evaluate the impact of treatment on level of inferior vena cava (IVC) thrombus.

V. To compare accruing center identified iRECIST progression and centrally identified iRECIST progression events on computed tomography (CT).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive one of the following immunotherapy regimens per physician discretion: nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes every 3 weeks for 4 doses followed by nivolumab IV over 30 minutes every 2 or 4 weeks; pembrolizumab IV over 30 minutes every 3 or 6 weeks and axitinib orally (PO) twice daily (BID); avelumab IV over 60 minutes every 2 weeks and axitinib PO BID; nivolumab IV over 30 minutes every 2 or 4 weeks and cabozantinib PO once daily (QD); OR pembrolizumab IV over 30 minutes every 3 or 6 weeks and lenvatinib PO QD. Treatment with immunotherapy continues in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) throughout the trial. Patients may also undergo a bone scan as clinically indicated and blood sample collection throughout the trial.

ARM II: Patients undergo SABR on 3 different days over 1-3 weeks and receive immunotherapy as in Arm I. Patients also undergo CT scan or MRI throughout the trial. Patients may also undergo a bone scan as clinically indicated and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 5 years, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of renal cell carcinoma prior to registration
* Node-positive unresectable (TxN1Mx) or metastatic (TxNxM1) based on the following diagnostic workup:

  * History/physical examination within 45 days prior to registration
  * CT/magnetic resonance imaging (MRI) of the chest/abdomen/pelvis within 45 days prior to registration
* Patients must have IMDC intermediate (1-2 factors) or poor risk disease (>= 3 factors)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with measurable disease (node positive or metastatic) as defined by RECIST version 1.1 excluding the primary renal tumor
* Patient not recommended for or refused immediate cytoreductive nephrectomy
* Candidate for standard of care therapy with either immuno-oncology (IO)-IO or IO-VEGF combination regimen
* Primary renal tumor measuring 20 cm or less in anterior to posterior dimension only on axial imaging
* Age >= 18
* Karnofsky performance status >= 60 within 45 days prior to registration
* Hemoglobin >= 8 g/dL (transfusions are allowed) (within 45 days prior to registration)
* Platelet count >= 50,000/mm^3 (within 45 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 45 days prior to registration)
* Calculated (Calc.) creatinine clearance >= 30 mL/min (within 45 days prior to registration)

  * Creatinine clearance (CrCl) >= 30 mL/min estimated by Cockcroft-Gault Equation
  * For African American patients specifically whose renal function is not considered adequate by the formula above, an alternative formula that takes race into account (Chronic Kidney Disease Epidemiology Collaboration CKD-EPI formula) should be used for calculating the related estimated glomerular filtration rate (GFR) with a correction factor for African American race creatinine clearance for trial eligibility, where GFR >= 30 mL/min/1.73m^2 will be considered adequate
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) (within 45 days prior to registration)
* Aspartate aminotransferase and alanine aminotransferase (AST and ALT) =< 3 x upper limit of normal (ULN) or < 5 x ULN if hepatic metastases present (within 45 days prior to registration)
* Patients with known human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Testing is not required for entry into protocol
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* The patient must agree to use a highly effective contraception, including men with vasectomies if they are having sex with a woman of childbearing potential or with a woman who is pregnant, while on study drug and for 6 months following the last dose of study drug. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Patients with planned treatment of all metastatic disease with definitive therapy including either surgery, ablative (non-palliative) doses of radiation, or intervention of some type (definitive interventional radiology techniques) to ALL metastatic sites rendering the patient without extra-renal measurable disease. Patients NOT planned for definitive treatment of all metastatic sites are eligible. Lesions radiated palliatively are not eligible for response assessment
* Patients with untreated or unstable brain metastases or cranial epidural disease

  * Note: Patients who have been adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks prior to registration as documented by MRI or CT imaging or deemed stable by clinical investigator are eligible. Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 4 weeks prior to registration as documented by MRI or CT imaging or deemed stable by clinical investigator
* Prior radiotherapy to the kidney that would result in overlap of radiation therapy fields treatment of the primary tumor
* Any systemic therapy for metastatic renal cell carcinoma (RCC) that was initiated > 90 days before registration, note that prior chemotherapy for a different cancer is allowed (completed > 3 years prior to registration)
* Severe, active comorbidity defined as follows:

  * Active autoimmune disease requiring ongoing therapy including systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications daily. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
  * History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies
  * Active tuberculosis (purified protein derivative [PPD] response without active tuberculosis [TB] is allowed)
  * Uncontrolled hypertension (systolic blood pressure [BP] >= 190 mmHg or diastolic BP > 110 mmHg)
  * Major surgery requiring hospital admission =< 28 days prior to registration
  * Any serious (requiring hospital stay or long term rehab) non-healing wound, ulcer, or bone fracture within 45 days prior to registration
  * Any arterial thrombotic (ST elevation myocardial infarction [STEMI], non-ST elevation myocardial infarction [NSTEMI], cerebrovascular accident [CVA], etc) events within 180 days prior to registration
  * Active New York (NY) Heart Association class 3-4 heart failure symptoms
  * Moderate or severe hepatic impairment (Child-Pugh B or C)
  * Any history of untreated pulmonary embolism or deep venous thrombosis (DVT) within 180 days prior to registration. (Any asymptomatic or treated pulmonary embolism or asymptomatic treated deep venous thrombosis > 30 days prior to registration is allowed)
  * Unstable cardiac arrhythmia within 180 days prior to registration
  * History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, bowel obstruction, or gastric outlet obstruction within 180 days prior to registration
  * History of or active inflammatory bowel disease
  * Malabsorption syndrome within 45 days prior to registration
* Pregnancy and individuals unwilling to discontinue nursing. For women of child bearing potential must have a negative pregnancy test =< 45 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Nephrectomy and radiographic progression-free survival (nrPFS) | From randomization to last follow-up, up to 8 years
  Nephrectomy and radiographic progression-free survival time is defined as time from randomization to the date of first radiographic progression, nephrectomy, death, or last negative evaluation (censored). nrPFS rates are estimated using the Kaplan-Meier method. Progression is determined by the Response Evaluation Criteria in Solid Tumors version 1.1 criteria modified for immunotherapy trials (iRECIST).

SECONDARY OUTCOMES:
Percentage of participants with complete or partial response | From randomization to disease progression
  Best overall response is determined by the iRECIST version 1.1.
Percentage of participants with complete or partial response in the primary renal mass | From randomization to disease progression
  Best overall response is determined by the iRECIST version 1.1.
Radiographic progression-free survival (rPFS) | From randomization to last follow-up, up to 8 years
  Radiographic progression-free survival time is defined as time from randomization to the date of first radiographic progression, death, or last negative evaluation (censored). rPFS rates are estimated using the Kaplan-Meier method. Radiographic progression is determined by the iRECIST version 1.1.
Nephrectomy and radiographic progression-free survival excluding nephrectomies that were performed for non-protocol specified reasons (nrPFS2) | From randomization to last follow-up, up to 8 years
  Nephrectomy and radiographic progression-free survival time (excluding nephrectomies that were performed for non-protocol specified reasons) is defined as time from randomization to the date of first radiographic progression, nephrectomy performed for protocol-stated reasons, death, or last negative evaluation (censored). nrPFS2 rates are estimated using the Kaplan-Meier method. Progression is determined by the iRECIST version 1.1.
Overall survival | From randomization to last follow-up, up to 8 years
  Overall survival time is defined as time from randomization to the date of death or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method.
Second-line therapy-free survival | From randomization to last follow-up, up to 8 years
  Second-line therapy-free survival time is defined as time from randomization to the date of the initiation of second-line therapy, death, or last known follow-up (censored). Second-line therapy-free survival rates are estimated using the Kaplan-Meier method.
Percentage of participants who undergo cytoreductive nephrectomy | From randomization to last follow-up, up to 8 years
Treatment-free survival | From randomization to last follow-up, up to 8 years
  Treatment-free survival time is defined as time from the discontinuation of protocol therapy to the date of death or last follow-up (censored). Treatment-free survival rates are estimated using the Kaplan-Meier method.
Percentage of participants with grade 3+ and with grade 4+ treatment-related adverse events | From randomization to last follow-up, up to 8 years
  Common Terminology Criteria for Adverse Events 5.0 grades adverse event severity from 1=mild to 5=death. Adverse events recorded as possibly, probably, or definitely related to protocol treatment will be considered to be treatment-related.

OTHER OUTCOMES:
nrPFS and overall survival | From randomization to last follow-up, up to 8 years
  Exploratory analyses will compare nrPFS and overall survival in four pre-defined subgroups: clear cell versus (vs.) non-clear cell histology, intermediate vs. poor International Metastatic RCC database consortium risk group, treatment with immuno-oncology (IO)-IO vs. IO-vascular endothelial growth factor, and sarcomatoid vs. non sarcomatoid variant. Forest plots will be constructed showing estimated hazard ratios from Cox models and 90% confidence intervals generated within each subgroup. Treatment-by-subgroup interaction terms will be incorporated into the Cox modelling to assess whether the effect of stereotactic ablative radiotherapy (SABR) varies significantly by subgroup; however, these analyses will be considered hypothesis-generating only.
Prognostic and predictive biomarkers | From randomization to last follow-up, up to 8 years
  Will be accomplished by including the biomarkers in Cox time-to-event regression models for the evaluation of prognostic factors. Treatment-by-biomarker interaction terms will be incorporated into the modelling process to assess for potential predictive markers.
Abscopal effect of SABR with systemic therapy | From randomization to disease progression
  These analyses will include only patients in the control arm who have not received any palliative radiation therapy and those in the experimental arm who have received protocol defined stereotactic body radiation therapy only without additional radiation therapy. Response rates among lesions outside the renal mass will be determined based in iRECIST criteria and compared using a chi-square test.
Impact of treatment on the level of inferior vena cava (IVC) thrombus | From randomization to last follow-up, up to 8 years
  Will be assessed by comparing the rates of IVC thromboembolism using Fisher's exact test. Cumulative incidence curves with death as a competing risk will also be generated and compared using the Fine-Gray test.
Accuracy of accruing center radiologist defined progression as compared with central radiology defined progression | From randomization to last follow-up, up to 8 years
  This will take place at the conclusion of the trial by our diagnostic radiologists. Will determine the number and proportion of center radiologist defined progressions (confirmed per iRECIST) that are validated/not validated upon central review. Will also examine all center radiologist defined pseudo progressions (i.e., not confirmed per iRECIST) and determine the number that are also declared pseudo progressions upon central review.

CONTACTS AND LOCATIONS:
Overall Officials: William A Hall, Principal Investigator — NRG Oncology
Locations (313):
- United States (308):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mills Health Center, San Mateo, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (2):
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- Ireland (2):
  - Beacon Hospital, Dublin, Co Dublin
  - Saint Lukes Hospital, Dublin, Co Dublin